CLINICAL TRIAL: NCT03450395
Title: The Effect of Oats Containing 1.4g Beta Glucan on Fecal Bacterial Population(s) and Plasma Cholesterol in Healthy Adults With Elevated Cholesterol Levels: a Randomized, Single-blind, Placebo-controlled, Cross-over Study
Brief Title: The Effect of Oats Containing 1.4g Beta Glucan on Fecal Bacterial Population(s) and Plasma Cholesterol in Healthy Adults With Elevated Cholesterol Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1720
Record Dates: First submitted 2018-01-29; First posted 2018-03-01 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Microbiome; Plasma Cholesterol; Prebiotic

STUDY DESIGN:
Intervention Model Description: For each of the two periods, a hot breakfast cereal will be consumed once daily for a duration of 6 weeks each. There will be a 4 week washout period in between each test substance.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cereal - Cream of Rice (Placebo Comparator): 40 g cream of rice
  Interventions: Other: Hot Cereal
- Cereal - Oats containing beta-glucan (Experimental): 40 g oats
  Interventions: Other: Hot Cereal

INTERVENTIONS:
Other: Hot Cereal — Intervention involves consumption of one hot cereal in the beginning of each day

SUMMARY:
The objectives of this study are to examine fecal bacterial population(s) and plasma cholesterol levels elicited by 40g of Oats and Cream of Rice over 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has given written informed consent;
2. Be between 18 and 65 years of age;
3. Has a BMI of between 18.5 - 30 Kg/m2;
4. Has a stable body weight (< 5% change) over the past 3-months;
5. Have elevated cholesterol levels, with a total cholesterol level >5.5mmol/L and <7mmol/L; and LDL cholesterol level ≥3.4 mmol/L and ≤4.9 mmol/L.
6. Is in general good health, as determined by the investigator;
7. Consumes a low to moderate fiber diet (9.9 - 25.1 g/day in males; 8.2 - 20.3 g/day in females);
8. Regularly consumes breakfast;
9. Avoid consuming prebiotic, probiotic or fiber rich supplements within 3 weeks prior to baseline visit, until the end of the study;
10. Avoid consumption of any whole grain oat products, within 3 weeks prior to baseline visit, until the end of the study;
11. Agrees to continue to consume the same dose of vitamin and/or mineral supplements, if applicable, for the duration of the study;
12. Maintain current level of physical activity;
13. Agree to keep detailed dietary and stool records;
14. Willing to consume the investigational products daily for the duration of the study.
15. Subject must have access to a microwave oven

Exclusion Criteria:

1. Females are pregnant, lactating or wish to become pregnant during the study. Female subject is currently either of:

   * non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or any female who is surgically sterilized (via documented hysterectomy or bilateral tubal ligation). (For purposes of this study, postmenopausal is defined as one year without menses), OR
   * child bearing potential, the subject is eligible to enter and participate in this study if she is not lactating and has a negative urine pregnancy test at the screening visit, visit 2 and upon completion of the study at visit 7. The subject must also agree to one of the following methods of contraception: i. Complete abstinence from intercourse two weeks prior to administration of study drug, throughout the clinical trial, until the completion of follow-up procedures or for two weeks following discontinuation of the study medication in cases where subject discontinues the study prematurely. (Subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent in the preceding 2 weeks when they present to the clinic for the Final Visit.) or, ii. has a male sexual partner who is surgically sterilized prior to the Screen Visit and is the only male sexual partner for that subject or, iii. sexual partner(s) is/are exclusively female or, iv. Oral contraceptives (either combined or progestogen only) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm. (Women of child-bearing potential using an oral contraceptive in combination with a double-barrier method of contraception are required to continue to use this form of contraception for 1 week following discontinuation of study medication).

     v. Use of double-barrier contraception, specifically, a spermicide plus a mechanical barrier (e.g. male condom, female diaphragm). The subject must be using this method for at least 1 week following the end of the study or, vi. Use of any intrauterine device (IUD) or contraceptive implant with published data showing that the highest expected failure rate is less than 1% per year. The subject must have the device inserted at least 2 weeks prior to the first Screen Visit, throughout the study, and 2 weeks following the end of the study,
2. Are hypersensitive to any of the components of the test products;
3. Is Coeliac, or has an intolerance to gluten;
4. Has taken antibiotics within the previous 3 months;
5. Has a history of drug and/or alcohol abuse at the time of enrolment;
6. Consumes greater than 2 servings/day of alcohol (e.g. >28 g ethanol/day);
7. Is a smoker;
8. Has a fasting blood glucose level outside the range of 3.0 - 6.0 mmol/L;
9. Has uncontrolled hypertension (systolic blood pressure ≥159 mm Hg or diastolic blood pressure ≥99 mm Hg);
10. Has made any major dietary changes in the past 3 months;
11. Planned major changes in life style (i.e. diet, dieting, exercise level, travelling) during the duration of the study;
12. Has a diagnosed eating disorder;
13. Is vegetarian/vegan diet or has food allergies or other issues with foods that would preclude intake of the study products;
14. Taking a medication/supplement that the investigator believes would impart or treat constipation, including iron, Imodium, Colon Clean, chronic or regular laxatives use or dependency on laxatives; and fiber supplements, within 3 weeks prior to baseline visit, until the end of the study;
15. Has an active gastrointestinal disorder or previous gastrointestinal surgery, other than an appendectomy
16. If taking chronic medications (e.g., hypertensive medications), they must have been taking the product for at least two months prior to screening and agree to maintain the same dosage throughout the study;
17. Subject is on any medication that has an effect on lowering cholesterol, such as use of beta blockers to treat hypertension or anxiety;
18. Has a metabolic or gastrointestinal diseases (i.e., diarrhea, Crohn's disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers, diabetes, hepatitis, HIV, cancer, etc.), with a history of such diseases;
19. Has a condition or taking a medication that the investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results; to include Statins (including atorvastatin (Lipitor and Torvast), fluvastatin (Lescol), lovastatin (Mevacor, Altocor, Altoprev), pitavastatin (Livalo, Pitava), pravastatin (Pravachol, Selektine, Lipostat), rosuvastatin (Crestor) and simvastatin (Zocor, Lipex)), Cholesterol Absorption Inhibitors (including Zetia (ezetimibe)), Niacin (nicotinic acid), Fibric acid derivatives (including Atromid-S (clofibrate), Lopid (gemfibrozil), and Tricor (fenofibrate)), Bile Acid Sequestrants (including cholestyramine, sold under the brand names Questran, Prevalite, and LoCholest, and colestipol (Colestid)) and Non Steroidal Anti-Inflammatory Drugs (NSAIDs), or have taken them in the past 28 days;
20. Taking a cholesterol lowering supplement, including, example Plant sterols/stanols, Fish Oil supplements, vitamin B supplements (e.g. Niacin and Niacinamide), red rice yeast extract, oat beta glucan, pharmaceutical garlic or have taken them in the past month;
21. Are severely immunocompromised (HIV positive, transplant patient, on antirejection medications, on a steroid for >30 days, or chemotherapy or radiotherapy within the last year);
22. Experiences alarm features such as weight loss, rectal bleeding, recent change in bowel habit (<3 months) or abdominal pain;
23. Have a malignant disease or any concomitant end-stage organ disease;
24. Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the trial;
25. Subjects may not be receiving treatment involving experimental drugs. If the subject has been in a recent experimental trial, these must have been completed not less than 60 days prior to this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

PRIMARY OUTCOMES:
Fecal bacterial population(s) | Baseline and Week 6
  Increase/decrease in desirable fecal bacterial groups (specifically, but not limited to, Bifidobacterium spp. and Lactobacillus/Enterococcus spp.).

SECONDARY OUTCOMES:
Fecal Bile Salt Hydrolase | Change from baseline and Week 6
  (ng-μg/g)
Fecal bile acid profile | Change from baseline Week 6
  (ng-μg/g)
Fecal bacterial diversity change | Change from baseline to Week 6
  Increase/decrease in desirable fecal bacterial groups (specifically, but not limited to, Bifidobacterium spp. and Lactobacillus/Enterococcus spp.). Increase would be better.
Serum FGF-19 | Change from baseline to Week 6
  Fibroblast growth factor (pg/ml)
Plasma total Cholesterol | Change from baseline to Week 6
  mmol/L, lower would be better
Change in Plasma HDL Cholesterol | Change from baseline to Week 6
  mmol/L, higher would be better
Change in Plasma LDL Cholesterol | Change from baseline to Week 6
  mmol/L, lower would be better
Change in Plasma Triglycerides | Change from baseline to Week 6
  mmol/L lower would be better
Change in Plasma Propionate (propanoic acid) | Change from baseline to Week 6
  (µM)
Stool frequency | Changes from baseline through 6 weeks
  Bowel movements recorded in daily diary
Change in stool consistency | Changes from baseline through 6 weeks
  Bristol Stool Scale, for each bowel movement, select closest appearance from chart. 7 types ranging from watery to hard lumps
Change in gastrointestinal symptoms | Changes from baseline through 6 weeks
  Pain, discomfort, bloating & flatulence recorded using subjective GI symptom ranking questionnaire 6 point scale from none to severe for 4 measures: pain, discomfort, bloating, flatulence. No changes would be better.
Quality of Life Score | Changes from baseline through 6 weeks
  SF-36 questionnaire (SF= Short form)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dinan, MD, PhD, Principal Investigator — Cork University Hospital & APC Microbiome Institute, University College Cork
Locations (1):
- Atlantia Food Clinical Trials, Cork, Ireland

IPD SHARING:
Plan to Share IPD: Undecided